CLINICAL TRIAL: NCT00313482
Title: A Phase II Trial of Docetaxel/Prednisone in Combination With Sargramostim as Treatment for Hormone-refractory Prostate Cancer
Brief Title: PII Trial of Docetaxel/Prednisone w/Sargramostim for HRPC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual
Sponsor: Veeda Oncology (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I-05-011
Record Dates: First submitted 2006-04-10; First posted 2006-04-12 (Estimated); Last update posted 2012-05-11 (Estimated); Status verified 2012-05

CONDITIONS: Hormone Refractory Prostate Cancer
MeSH Terms: interventions — sargramostim; Docetaxel; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Sargramostim — 250 mcg/m2 SC days 2-15 of each cycle
  Other Names: Leukine
Drug: Docetaxel — 75 mg/m2 IV over 1 hour on Day 1 of each cycle
  Other Names: Taxotere
Drug: Prednisone — 5 mg orally BID on Day 1 continuously

SUMMARY:
This is a Phase II, open-label study in male patients with metastatic HRPC.

Each cycle will be 21 days (3 weeks). Patients will receive the following drugs:

* Docetaxel 75 mg/m2 IV given over 1 hour on Day 1.
* Prednisone 5 mg orally twice daily beginning on Day 1 and continuing until disease progression.
* Sargramostim 250 mcg/m2 SC on Days 2-15 of each cycle. Patients will be evaluated every 4 cycles (12 weeks) for response using RECIST criteria. PSA response will be evaluated according to the National Cancer Institute (NCI) PSA Working Group Criteria. To evaluate the safety of this drug combination, patients will be evaluated at each clinic visit for adverse events. Toxicities will be assessed per National Cancer Institute (NCI) CTCAE Version 3.0.

Those patients achieving stable disease or better will continue therapy. Those patients experiencing progressive disease will be taken off study.

Patients will receive a maximum of 10 cycles of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have signed an IRB-approved informed consent.
2. Patients must be male with histologically confirmed metastatic adenocarcinoma of the prostate with progressive disease, despite androgen deprivation.
3. Patients must have a history of prior hormone therapy (must fulfill one of the following criteria):

   * Castration and/or luteinizing-hormone releasing hormone (LHRH) agonist
   * Antiandrogen therapy (flutamide, nilutamide, bicalutamide, or cyproterone acetate)
   * Antiandrogen therapy withdrawal
   * Estramustine monotherapy
   * Other hormonal therapy (eg, ketoconazole). Note: Patients must be off ketoconazole at least 1 month. If PSA is decreasing, the patient must demonstrate a rising PSA on at least 2 sequential reading at least 2 weeks apart.
4. Patients must have a serum testosterone <50 ng/dL (if the patient has not undergone orchiectomy, he must continue primary androgen deprivation with LHRH analogue).
5. Patient must fulfill one of the following criteria:

   * Patients with measurable disease:

   Patients must have disease progression defined by the RECIST criteria.
   * Patients with no measurable disease:

   Patients with PSA only disease must have an elevated PSA by Consensus Criteria. -OR-
   * Patients with a positive bone scan must also have elevated PSA defined by Consensus Criteria.
6. Progressive disease (as defined above) must be documented after discontinuation of hormonal therapy.
7. Patients who are receiving an antiandrogen as part of primary androgen ablation must also demonstrate disease progression following discontinuation of the antiandrogen.
8. Patients on antiandrogen therapy must discontinue therapy and subsequently demonstrate disease progression (at least 4 weeks since prior flutamide or nilutamide, 8 weeks since prior bicalutamide).
9. Patients must have discontinued all agents or herbal products known to decrease PSA levels (eg, Megace [megestrol acetate], Saw Palmetto, and PC-SPEC) or any systemic corticosteroid at least 4 weeks prior to enrollment.
10. Patients must have Karnofsky Performance Status (PS) >60.
11. Patients must have a life expectancy >3 months.
12. Patients must be >18 years of age.
13. Patients may have received prior radiation (except for radiation to the entire pelvis), provided that less than 25% of the bone marrow has been treated, and the patient has recovered from the acute toxic effects of treatment prior to trial enrollment. Irradiation of a symptomatic lesion, or one that may produce disability (eg, unstable femur) prior to study initiation is permitted, provided other measurable disease is present. Prior radiation treatment must have been completed at least 4 weeks prior to enrollment. Lesions that have been irradiated in the advanced disease setting may not be included as sites of measurable disease.
14. Patients must agree to use effective contraceptive measures during study treatment and for a reasonable time thereafter.
15. Patients must have absolute neutrophil count (ANC) >1500/μL, platelet count >100,000/μL, and hemoglobin >8 mg/dL.
16. Patients must have alanine transaminase (ALT), aspartate transaminase (AST), and total bilirubin within normal limits (WNL), serum creatinine <1.5 x upper limit of normal (ULN).
17. Patients must be willing and able to self-administer or have a caregiver who can administer in compliance with the protocol (sargramostim).

Exclusion Criteria:

1. Prior systemic chemotherapy for the treatment of HRPC, with the exception of estramustine monotherapy.
2. Prior treatment with ketoconazole, aminoglutethimide, or corticosteroids for the treatment of progressive prostate cancer.
3. No prior immunotherapy with the exception of routine immunizations.
4. Myocardial infarction or significant change in anginal pattern within the last 6 months, symptomatic congestive heart failure (New York Heart Association Class III or higher, see Appendix II) or uncontrolled cardiac arrhythmia.
5. Patients with known HIV-positive status.
6. Major surgery or radiation therapy <4 weeks prior to enrollment.
7. Prior radiopharmaceuticals (strontium, samarium) within 8 weeks prior to enrollment.
8. Patients with a history of severe hypersensitivity reaction to docetaxel, prednisone, sargramostim, yeast-derived products, other drugs formulated with polysorbate 80, or any of the components in these drugs.
9. Patients with poorly controlled diabetes (fasting blood glucose >250 mg/dL) despite optimization of medical therapy.
10. Patients with serious uncontrolled intercurrent infections, nonmalignant medical illnesses, or active uncontrolled autoimmune disease. Note: suppressive antibiotic therapy for chronic urinary tract infections is allowed.
11. Patients with a systemic fungal infection.
12. Patients with psychiatric illness/social situations that would limit compliance with treatment or adequate informed consent.
13. Any patient who is unable to comply with requirements of study.
14. Patients with symptomatic peripheral neuropathy Grade >2 (NCI Common Toxicity Criteria Version 3.0.
15. Patients with known brain or leptomeningeal involvement.
16. Patients with second primary malignancy, except adequately treated nonmelanomatous carcinoma of the skin or other malignancy treated >5 years previously and with no other evidence of recurrence.

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2006-04; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the effects of the combination of docetaxel/prednisone with sargramostim on progression-free survival in chemotherapy-naïve male patients with hormone-refractory prostate cancer (HRPC). | unk

SECONDARY OUTCOMES:
To evaluate the response (as demonstrated by PSA and/or measurable disease) to the combination of docetaxel/prednisone with sargramostim. | unk
To evaluate the 1-year and 2-year survival following treatment with the combination of docetaxel/prednisone with sargramostim. | unk
To evaluate the safety of the combination of docetaxel/prednisone with sargramostim. | unk

CONTACTS AND LOCATIONS:
Overall Officials: Evan R Berger, MD, Principal Investigator — North Shore Hematology Oncology Associates
Locations (1):
- Veeda Oncology, Columbus, Ohio, United States